CLINICAL TRIAL: NCT01807325
Title: RNA Sequencing of Solid and Cystic Lesions of the Pancreas
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Providence Health & Services (Other)
Responsible Party: Sponsor
Other Study IDs: IRB8317
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Pancreas Cyst; Pancreas Mass
MeSH Terms: conditions — Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pancreas biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pancreas cysts and solid masses: patents referred for solid and cystic lesions of the pancreas who will have a biopsy for usual medical care.
  Interventions: Procedure: pancreas biopsy

INTERVENTIONS:
Procedure: pancreas biopsy — patients who are already having a pancreas biopsy will be invited to enroll. After obtaining enough tissue for usual medical care, we will divert some tissue for the study.
  Other Names: RNA sequencing of pancreas tissue

SUMMARY:
The nature of cysts and solid masses in the pancreas can be difficult to diagnose. They may be benign, precancerous, or cancer. Current tests such as cytology (looking under a microscope) and tumor markers do not always give us the answer. The investigators are looking for genetic markers on biopsy specimens from the pancreas that will give us a better test for diagnosis. This study is only for diagnosing these lesions. The investigators are not treating any patients.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years old,
* not pregnant,
* referred for endoscopic ultrasound,
* have a cyst or mass of the pancreas needing diagnosis.

Exclusion Criteria:

* pregnant,
* less than age 18,
* no mass or cyst found.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult, nonpregnant patients referred for endoscopic ultrasound to evaluate solid or cystic lesion of the pancreas.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Gene classifier that will classify lesions as benign or malignant with 95% certainty | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rodriguez, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Providence St Vincent Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon